CLINICAL TRIAL: NCT06131463
Title: Assessing the Impact of Using the Electrocardiogram Function in Smart Watches on the Level of Anxiety (GAD-7) Among University Students and Employees
Brief Title: Anxiety Associated With the Use of the Electrocardiogram Function in Smart Watches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ITMO University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: be-healthy-smart-watches
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Wellness 1; Anxiety Disorders; Depression
Keywords: Anxiety; Depression; ECG; Smartwatch; Randomized trial
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Electrocardiography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECG function is enabled (Experimental): Electrocardiogram (ECG) feature on the smartwatch is enabled
  Interventions: Device: Electrocardiogram (ECG) feature in smart watches
- ECG function is not enabled (No Intervention): Electrocardiogram (ECG) feature on the smartwatch is not enabled

INTERVENTIONS:
Device: Electrocardiogram (ECG) feature in smart watches — A study participant that is randomly assigned to the experimental group should enable the ECG function on his or her smart watch and make sure that there is synchronization with a corresponding application on his or her mobile phone. The ECG function must stay enabled, and the participant should wear the smartwatch every day for 30 days.
  Arms: ECG function is enabled

SUMMARY:
The integration of electrocardiography (ECG) functionality into smartwatches is primarily intended to screen for atrial fibrillation, a frequent cause of ischemic stroke, among people aged 50 years and older. However, it should be noted that recommendations for atrial fibrillation screening are controversial, and several organizations and communities do not recommend screening outside of at-risk groups.

Some smart device manufacturers do not recommend using the ECG function for anyone under the age of 22. However, young people are frequent users of wearable devices. One of the most common cardiologic diseases at the age of 18-30 is benign heart rhythm disorder, which often does not require diagnosis or treatment and can be considered normal.

That said, notification of the detection of atrial fibrillation can affect psycho-emotional well-being, particularly anxiety.

This study will assess the level of psycho-emotional health (anxiety level) of the study participants. Participant observation will provide an opportunity to identify associations between the use of the ECG recording function on wearable devices and levels of anxiety and depression. It is hypothesized that the use of smartwatches with the ECG function activated will not lead to a change in anxiety levels on the GAD-7 scale among the study participants. This assumes that after 30 days of use, the mean value of the GAD-7 scale in the intervention group and the control group will be the same.

ELIGIBILITY:
Inclusion Criteria:

* Status of a student or employee of ITMO University;
* Availability of a smart watch with ECG function (Apple Watch Series 4 and newer, Galaxy Watch Active2, Samsung Galaxy Watch Series 3 and newer or similar with ECG function);
* Availability of a Galaxy smartphone running Android 7.0 or newer or availability of an iPhone 8 and newer smartphone with the latest version of iOS.
* Signed Informed consent and Consent for Data Processing of Personal Data;
* Absence of previously diagnosed clinically significant cardiovascular pathology.

Exclusion Criteria:

* Participants under the age of 22 cannot be included in the study;
* Participants in the acute phase of any disease or in the exacerbation of chronic diseases are excluded from the study.

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Anxiety level | 30 days
  Anxiety level is measured 30 days after the enrolment with Generalized Anxiety Disorder 7-item (GAD-7) which is a tool based on seven items which are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.

SECONDARY OUTCOMES:
Depression | 30 days
  Depression is assessed 30 days after the enrolment with Patient Health Questionnaire-9 (PHQ-9) that can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Depression | 90 days
  Depression is assessed 90 days after the enrolment with Patient Health Questionnaire-9 (PHQ-9) that can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Anxiety level | 90 days
  Anxiety level is measured 90 days after the enrolment with Generalized Anxiety Disorder 7-item (GAD-7) which is a tool based on seven items which are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Heart rhythm disturbances | 90 days
  The frequency of detection of clinically significant and clinically insignificant heart rhythm disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Liubov Maliugina, MD, Principal Investigator — ITMO University
Locations (1):
- ITMO University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tison GH, Sanchez JM, Ballinger B, Singh A, Olgin JE, Pletcher MJ, Vittinghoff E, Lee ES, Fan SM, Gladstone RA, Mikell C, Sohoni N, Hsieh J, Marcus GM. Passive Detection of Atrial Fibrillation Using a Commercially Available Smartwatch. JAMA Cardiol. 2018 May 1;3(5):409-416. doi: 10.1001/jamacardio.2018.0136. PMID 29562087
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] US Preventive Services Task Force; Davidson KW, Barry MJ, Mangione CM, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Epling JW Jr, Kubik M, Li L, Ogedegbe G, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Atrial Fibrillation: US Preventive Services Task Force Recommendation Statement. JAMA. 2022 Jan 25;327(4):360-367. doi: 10.1001/jama.2021.23732. PMID 35076659
- [Background] Rosman L, Gehi A, Lampert R. When smartwatches contribute to health anxiety in patients with atrial fibrillation. Cardiovasc Digit Health J. 2020 Jul-Aug;1(1):9-10. doi: 10.1016/j.cvdhj.2020.06.004. Epub 2020 Aug 28. No abstract available. PMID 34386784
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Toussaint A, Husing P, Gumz A, Wingenfeld K, Harter M, Schramm E, Lowe B. Sensitivity to change and minimal clinically important difference of the 7-item Generalized Anxiety Disorder Questionnaire (GAD-7). J Affect Disord. 2020 Mar 15;265:395-401. doi: 10.1016/j.jad.2020.01.032. Epub 2020 Jan 15. PMID 32090765
- See also: How to use the ECG app on Apple Devices — https://support.apple.com/en-us/HT208955